CLINICAL TRIAL: NCT02807116
Title: A Phase 1, Open-Label, Drug-Interaction Study to Evaluate the Effect of Rifampin, a Potent CYP3A4 Inducer, on the Systemic Exposure of Pacritinib in Healthy Subjects
Brief Title: Drug-Interaction Study to Evaluate the Effect of Rifampin, a Potent CYP3A4 Inducer, on the Systemic Exposure of Pacritinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PAC106
Record Dates: First submitted 2016-05-03; First posted 2016-06-21 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2016-06

CONDITIONS: Healthy Subjects
Keywords: Drug-Interaction Study
MeSH Terms: interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Rifampin

ARMS (1):
- Pacritinib and Rifampin (Experimental): On Day 1, subjects received a single oral 400-mg dose of pacritinib. On Days 8 through 17, following a 7-day washout period, 600-mg oral doses of rifampin were administered QD. It was anticipated that steady-state concentrations of rifampin would be achieved by Day 17. On Day 17, a single oral 400-mg dose of pacritinib was co-administered with the final 600-mg dose of rifampin.
  Interventions: Drug: Pacritinib; Drug: Rifampin; Drug: Pacritinib and Rifampin

INTERVENTIONS:
Drug: Pacritinib — Subjects received a single oral 400-mg dose of pacritinib
  Other Names: PAC400 mg
Drug: Rifampin — Subjects received 600-mg oral doses of rifampin; administered QD following a 7-day washout period
  Other Names: Rifampin600 mg
Drug: Pacritinib and Rifampin — On Day 17, a single oral 400-mg dose of pacritinib was co-administered with the final 600-mg dose of rifampin.
  Other Names: PAC400 mg and rifampin 600mg

SUMMARY:
The primary objective is to evaluate the effect of rifampin, a potent cytochrome P450 3A4 inducer, at steady-state on the systemic exposure of a single dose of pacritinib in healthy subjects.

DETAILED DESCRIPTION:
This was a single-center, open-label, one-way crossover, drug-interaction study. On Day 1, subjects received a single oral 400-mg dose of pacritinib. Following a 7-day washout period, 600-mg oral doses of rifampin were administered once daily (QD) on Days 8 through 17. It was anticipated that steady-state concentrations of rifampin would be achieved by Day 17. On Day 17, a single oral 400-mg dose of pacritinib was co-administered with the final 600-mg dose of rifampin.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria may be included in the study:

1. males or females, between 18 and 55 years of age, inclusive;
2. BMI between 18.5 and 32.0 kg/m2, inclusive;
3. in good health, determined by no clinically significant findings from medical history, physical examination, and vital sign measurements;
4. clinical laboratory evaluations (including clinical chemistry panel [fasted at least 10 hours], CBC, and UA) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator and in consultation with the Sponsor;
5. negative test for selected drugs of abuse (including alcohol) at Screening and at Check-in (Day -1);
6. negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV]) and negative HIV antibody screens;
7. females of childbearing potential must be non-pregnant and non-lactating, and agree to use one of the following forms of contraception from the time of signing the Informed Consent Form (ICF) or 10 days prior to Check-in (Day -1) until 30 days after the final dose administration: non-hormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; intravaginal system (eg, NuvaRing®); diaphragm with spermicide; cervical cap with spermicide; male sexual partner who agrees to use a male condom with spermicide; sterile sexual partner; or abstinence. Oral, implantable, transdermal, or injectable hormonal contraceptives may not be used from the time of signing the ICF or 10 days prior to Check-in (Day -1) until 14 days after the final dose administration. For all females, the pregnancy test result must be negative at Screening and Check-in (Day -1). Females not of childbearing potential must have had continuous amenorrhea for at least 12 months or surgically sterile (eg, tubal ligation, hysterectomy) for at least 90 days prior to Screening;
8. males will either be surgically sterile (ie, vasectomy, documented in the medical record by a physician) or agree to use, from Check-in (Day -1) until 90 days following Study Completion/Early Termination (ET), one of the following approved methods of contraception: male condom with spermicide; sterile sexual partner; or use by female sexual partner of an IUD with spermicide; a female condom with spermicide; a contraceptive sponge with spermicide; an intravaginal system; a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives. Subjects must agree to refrain from sperm donation from Check-in (Day -1) until 90 days following Study Completion/ET;
9. able to comprehend and willing to sign an ICF

Exclusion Criteria:

The following will exclude potential subjects from the study:

1. history or clinical manifestation of clinically significant cardiovascular, pulmonary, hepatic (eg, hepatitis), renal, hematologic, gastrointestinal (eg, celiac disease, peptic ulcer, gastroesophageal reflux, inflammatory bowel disease), metabolic, allergic, dermatological, neurological, or psychiatric disorder (as determined by the Investigator; appendectomy and cholecystectomy are not considered to be clinically significant procedures);
2. abnormalities in liver function tests (any/all of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase > upper limit of normal [ULN]; gamma-glutamyl transferase > ULN; or total bilirubin

   > ULN) or kidney function tests (serum creatinine > ULN); laboratory values may be confirmed by repeat;
3. history of malignancy, except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps;
4. history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, including rifampin, unless approved by the Investigator in consultation with the Sponsor;
5. history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed;
6. history of Gilbert's Syndrome;
7. history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant; QT corrected for heart rate using Fridericia's formula (QTcF) >450 msec; or factors that increase risk for QTc interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome);
8. history of alcoholism or drug addiction within 1 year prior to Check-in (Day -1);
9. use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1) and during the entire study;
10. receipt of blood products within 2 months prior to Check-in (Day -1);
11. participation in any other investigational drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days prior to Check-in (Day -1), whichever is longer;
12. donation of blood from 30 days prior to Screening through Study Completion/ET, inclusive, or of plasma from 2 weeks prior to Screening through Study Completion/ET, inclusive;
13. use of any prescription medications and/or products within 14 days prior to Check-in (Day -1) and during the entire study, unless deemed acceptable by the Investigator in consultation with the Sponsor;
14. use of oral, implantable, injectable, or transdermal hormonal contraceptives within 10 days prior to Check-in (Day -1) or from the time of signing the ICF (females only) until 14 days after the final dose administration;
15. use of any over-the-counter, non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in (Day -1) and during the entire study, unless deemed acceptable by the Investigator;
16. consumption of alcohol- or caffeine-containing foods and beverages for 72 hours prior to Check-in (Day -1) and during the entire study;
17. consumption of grapefruit-containing foods and beverages or other CYP3A4 inhibitors or inducers for 72 hours prior to Check-in (Day -1) and during the entire study;
18. participation in strenuous exercise for 48 hours prior to Check-in (Day -1) and during the period of confinement at the CRU; subjects will otherwise maintain their normal level of physical activity throughout the entire study (ie, will not begin a new exercise program nor participate in any unusually strenuous physical exertion);
19. poor peripheral venous access;
20. any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Estimate ratios of geometric mean values and the corresponding 90% confidence intervals (CIs) for pacritinib treatments with and without rifampin | Approx. one month
  Estimate ratios of geometric mean values and the corresponding 90% confidence intervals (CIs) for pacritinib treatments with and without rifampin to assess the potential for clinical interaction with CYP3A4 inducers.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Day 1 to Day 24
  To compare the safety and tolerability of single doses of pacritinib alone and in the presence of steady-state rifampin in healthy subjects
The maximum plasma concentration (Cmax). | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule with or without rifampin in healthy subjects
The time to reach maximum plasma concentration (tmax) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule with or without rifampin in healthy subjects
The area under the plasma concentration-time curve from time zero to time of the last measured concentration above the limit of quantification (AUC0-t) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule with or without rifampin in healthy subjects
The area under the plasma concentration-time curve from zero to infinity (AUC0-∞) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule with or without rifampin in healthy subjects
The apparent terminal elimination rate constant (λZ) and the respective apparent terminal elimination half-life (t½) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule with or without rifampin in healthy subjects
The apparent volume of distribution (Vd) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule with or without rifampin in healthy subjects
The apparent total body clearance (CL/F) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  The following pharmacokinetic parameters of pacritinib and major human metabolites were assessed following 400 mg single-dose administration of pacritinib capsule with or without rifampin in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Hugh A Coleman, DO, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes